CLINICAL TRIAL: NCT05241457
Title: Achieving Meaningful Clinical Benchmarks With Ekso Gait Training During Acute Stroke Inpatient Rehabilitation.
Status: Recruiting | Type: Observational
Sponsor: Sunnyview Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Karah Lenge, Doctor of Physical Therapy, Sunnyview Rehabilitation Hospital
Other Study IDs: 21-1116-1
Record Dates: First submitted 2022-01-24; First posted 2022-02-15 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Stroke; Stroke, Acute; Cerebrovascular Accident; Cerebrovascular Accident, Acute
Keywords: Exoskeleton; Gait training; Inpatient rehabilitation; Ekso gait training
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Standard of care group: Patients will receive the standard physical therapy sessions that they would normally receive during their IRF stay, (60 to 90 min sessions, 5 to 6 days/week). This group will not receive Ekso exoskeleton gait training.
  Interventions: Procedure: Standard physical therapy
- Ekso exoskeleton gait training group: Patients in the Ekso group will have several (2 to 3) of their standard of care sessions replaced with Ekso gait training sessions each week.
  Interventions: Device: Ekso gait training; Procedure: Standard physical therapy

INTERVENTIONS:
Device: Ekso gait training — Ekso sessions will be 60 minutes each. Patients will be measured to optimize Ekso fit during their initial training session. Ekso settings will be progressed as deemed appropriate by the trained clinician. The progression of Ekso settings allows the patient to use their maximum effort while the Ekso assists only as much as the patient requires to complete stepping. Patients may also spend time working on pre-gait activities and balance activities including weight shifting, stepping in place, side-stepping and backwards ambulation based on the patient's needs as determined by the clinician.
  Groups: Ekso exoskeleton gait training group
Procedure: Standard physical therapy — Standard physical therapy sessions will be 60 to 90 minutes a day. Clinicians typically focus on gait, balance, and strengthening activities that address goals related to functional mobility. Other devices that would normally be used during PT sessions, including the Lite Gait and Rifton tram body weight support devices and electrical stimulation devices including the XCITE and RT300 (from Restorative Therapies).

SUMMARY:
The Ekso (Ekso Bionics) is a wearable exoskeleton that provides robotic support and walking assistance for patients with lower extremity paralysis. Research suggests that exoskeleton-assisted gait training is as effective as conventional gait training at improving walking outcomes and balance during both the chronic and subacute period following stroke (Goffredo et al., 2019; Molteni et al., 2017; Molteni et al., 2021; Nam et al., 2019; Rojek, 2019).

Exoskeleton-assisted gait training during acute inpatient rehabilitation provides a means for patients to actively participate in gait training during the early and most severe stages of stroke recovery. Most acute inpatient rehabilitation facilities (IRFs) report a feasibility of 5-8 Ekso sessions during inpatient stays and demonstrate significant improvement from baseline (Nolan et al., 2020; Swank, 2020). Nolan et al. (2020) demonstrated that stroke patients receiving Ekso ambulated 1640 feet more than patients undergoing more conventional gait training techniques during inpatient rehabilitation, suggesting that the exoskeleton may offer additional benefit during this phase of recovery. Despite promising evidence, there have been no randomized controlled trials within the IRF setting.

Because Ekso-gait training increases the number of steps patients can take, during acute inpatient physical therapy (PT), the investigators hypothesize that patients who participate in Ekso-gait training will demonstrate quicker improvements in balance, gait speed, endurance and independence in functional ambulation during their stay in the IRF.

In this study, eligible patients admitted to Sunnyview Rehabilitation Hospital (SRH) for rehabilitation following stroke will be randomized to receive conventional or Ekso-gait training therapy. Meaningful clinical benchmarks for balance and walking will be assessed using the Berg Balance Scale (BBS) (Alghadir, 2018; Moore, 2018), the 10 Meter Walk Test (10MWT) (Bowden, 2008; Moore, 2018), the Six Minute Walk Test (6MWT) (Kubo et al., 2020; Moore, 2018), and Functional Ambulation Category (FAC) (Mehrholz, 2007). Achieving these benchmark scores are associated with several positive outcomes, including increased ability to ambulate in the community and reduced risk of falling (Alghadir, 2018; Bowden, 2008; Kubo et al., 2020). The investigators also hypothesize that patients in the Ekso cohort will report greater value/usefulness when compared to patients receiving standard care.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient at Sunnyview Rehabilitation Hospital
* Right or left hemispheric stroke
* >18 years of age

Exclusion Criteria:

* No paresis
* Paraplegia
* Quadriplegia
* FAC of 2,3 or 4
* Weight > 220 lbs (Ekso manufacturer criteria)
* Height > 6'4" (Ekso manufacturer criteria)
* > 3 months post stroke onset
* Comorbidities affecting gait (LE fractures, Parkinson's, Severe Polyneuropathy)
* LE/sacral wounds that come into contact with the Ekso
* LE contractures that cannot be accommodated by Ekso
* Prior Stroke
* Weight Bearing Restrictions 8
* Unable to follow 1-2 step commands.
* Contact precautions for COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatient Rehabilitation Facility
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-03-11 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
10-meter walk test at self-selected speed (10MWT, SSS) | T1 (Day 14-16)
  Used to assess walking speed over a short distance at the patient's chosen speed.
10-meter walk test at self-selected speed (10MWT, SSS) | T2 (Day 20-22)
  Used to assess walking speed over a short distance at the patient's chosen speed.
10-meter walk test at self-selected speed (10MWT, SSS) | T3 (Day 27-29)
  Used to assess walking speed over a short distance at the patient's chosen speed.
10-meter walk test at fast speed (10MWT, fast) | T1 (Day 14-16)
  Used to assess walking speed over a short distance at a self-determined speed that is as fast as they can safely walk.
10-meter walk test at fast speed (10MWT, fast) | T2 (Day 20-22)
  Used to assess walking speed over a short distance at a self-determined speed that is as fast as they can safely walk.
10-meter walk test at fast speed (10MWT, fast) | T3 (Day 27-29)
  Used to assess walking speed over a short distance at a self-determined speed that is as fast as they can safely walk.
BERG Balance scale | T1 (Day 14-16)
  A 14-item scale used to assess sitting, standing, static and dynamic balance. The test focuses on the ability to maintain a position and adjust posture to complete functional movements.
BERG Balance scale | T2 (Day 20-22)
  A 14-item scale used to assess sitting, standing, static and dynamic balance. The test focuses on the ability to maintain a position and adjust posture to complete functional movements.
BERG Balance scale | T3 (Day 27-29)
  A 14-item scale used to assess sitting, standing, static and dynamic balance. The test focuses on the ability to maintain a position and adjust posture to complete functional movements.
6-minute walk test (6MWT) | T1 (Day 14-16)
  Used to assess walking endurance and aerobic capacity. The total distance a patient walks over six minutes is recorded.
6-minute walk test (6MWT) | T2 (Day 20-22)
  Used to assess walking endurance and aerobic capacity. The total distance a patient walks over six minutes is recorded.
6-minute walk test (6MWT) | T3 (Day 27-29)
  Used to assess walking endurance and aerobic capacity. The total distance a patient walks over six minutes is recorded.

SECONDARY OUTCOMES:
Functional Ambulation Category (FAC) | T1 (Day 14-16)
  A five-point scale used to categorize a patient's ambulation status, ranging from independent walking outside to non-functional walking.
Functional Ambulation Category (FAC) | T2 (Day 20-22)
  A five-point scale used to categorize a patient's ambulation status, ranging from independent walking outside to non-functional walking.
Functional Ambulation Category (FAC) | T3 (Day 27-29)
  A five-point scale used to categorize a patient's ambulation status, ranging from independent walking outside to non-functional walking.
Intrinsic Motivation Inventory (IMI) | T2 (Day 20-22)
  The value of the intervention as perceived by patients

CONTACTS AND LOCATIONS:
Overall Officials: Karah Lenge, DPT, Principal Investigator — Sunnyview Rehabilitation Hospital; Allison Tallon, DPT, Principal Investigator — Sunnyview Rehabilitation Hospital
Locations (1):
- Sunnyview, Schenectady, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alghadir AH, Al-Eisa ES, Anwer S, Sarkar B. Reliability, validity, and responsiveness of three scales for measuring balance in patients with chronic stroke. BMC Neurol. 2018 Sep 13;18(1):141. doi: 10.1186/s12883-018-1146-9. PMID 30213258
- [Background] Bowden MG, Balasubramanian CK, Behrman AL, Kautz SA. Validation of a speed-based classification system using quantitative measures of walking performance poststroke. Neurorehabil Neural Repair. 2008 Nov-Dec;22(6):672-5. doi: 10.1177/1545968308318837. PMID 18971382
- [Background] Goffredo M, Guanziroli E, Pournajaf S, Gaffuri M, Gasperini G, Filoni S, Baratta S, Damiani C, Franceschini M, Molteni F; Italian EksoGait Study Group. Overground wearable powered exoskeleton for gait training in subacute stroke subjects: clinical and gait assessments. Eur J Phys Rehabil Med. 2019 Dec;55(6):710-721. doi: 10.23736/S1973-9087.19.05574-6. Epub 2019 Feb 4. PMID 30723189
- [Background] Kubo H, Nozoe M, Kanai M, Furuichi A, Onishi A, Kajimoto K, Mase K, Shimada S. Reference value of 6-minute walk distance in patients with sub-acute stroke. Top Stroke Rehabil. 2020 Jul;27(5):337-343. doi: 10.1080/10749357.2019.1704372. Epub 2019 Dec 18. PMID 31851872
- [Background] Mehrholz J, Wagner K, Rutte K, Meissner D, Pohl M. Predictive validity and responsiveness of the functional ambulation category in hemiparetic patients after stroke. Arch Phys Med Rehabil. 2007 Oct;88(10):1314-9. doi: 10.1016/j.apmr.2007.06.764. PMID 17908575
- [Background] Molteni F, Gasperini G, Gaffuri M, Colombo M, Giovanzana C, Lorenzon C, Farina N, Cannaviello G, Scarano S, Proserpio D, Liberali D, Guanziroli E. Wearable robotic exoskeleton for overground gait training in sub-acute and chronic hemiparetic stroke patients: preliminary results. Eur J Phys Rehabil Med. 2017 Oct;53(5):676-684. doi: 10.23736/S1973-9087.17.04591-9. Epub 2017 Jan 24. PMID 28118698
- [Background] Molteni F, Guanziroli E, Goffredo M, Calabro RS, Pournajaf S, Gaffuri M, Gasperini G, Filoni S, Baratta S, Galafate D, Le Pera D, Bramanti P, Franceschini M, On Behalf Of Italian Eksogait Study Group. Gait Recovery with an Overground Powered Exoskeleton: A Randomized Controlled Trial on Subacute Stroke Subjects. Brain Sci. 2021 Jan 14;11(1):104. doi: 10.3390/brainsci11010104. PMID 33466749
- [Background] Moore JL, Potter K, Blankshain K, Kaplan SL, O'Dwyer LC, Sullivan JE. A Core Set of Outcome Measures for Adults With Neurologic Conditions Undergoing Rehabilitation: A CLINICAL PRACTICE GUIDELINE. J Neurol Phys Ther. 2018 Jul;42(3):174-220. doi: 10.1097/NPT.0000000000000229. PMID 29901487
- [Background] Nam YG, Lee JW, Park JW, Lee HJ, Nam KY, Park JH, Yu CS, Choi MR, Kwon BS. Effects of Electromechanical Exoskeleton-Assisted Gait Training on Walking Ability of Stroke Patients: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2019 Jan;100(1):26-31. doi: 10.1016/j.apmr.2018.06.020. Epub 2018 Jul 25. PMID 30055163
- [Background] Nolan KJ, Karunakaran KK, Chervin K, Monfett MR, Bapineedu RK, Jasey NN, Oh-Park M. Robotic Exoskeleton Gait Training During Acute Stroke Inpatient Rehabilitation. Front Neurorobot. 2020 Oct 30;14:581815. doi: 10.3389/fnbot.2020.581815. eCollection 2020. PMID 33192438
- [Background] Rojek A, Mika A, Oleksy L, Stolarczyk A, Kielnar R. Effects of Exoskeleton Gait Training on Balance, Load Distribution, and Functional Status in Stroke: A Randomized Controlled Trial. Front Neurol. 2020 Jan 15;10:1344. doi: 10.3389/fneur.2019.01344. eCollection 2019. PMID 32010039
- [Background] Swank C, Sikka S, Driver S, Bennett M, Callender L. Feasibility of integrating robotic exoskeleton gait training in inpatient rehabilitation. Disabil Rehabil Assist Technol. 2020 May;15(4):409-417. doi: 10.1080/17483107.2019.1587014. Epub 2019 Mar 19. PMID 30887864
- See also: Ekso Bionics - Exoskeleton device — https://eksobionics.com/